### STATISTICAL ANALYSIS PLAN

Study: EP0009

**Product: Lacosamide** 

A MULTICENTER, OPEN-LABEL, UNCONTROLLED, LONG-TERM, EXTENSION STUDY TO EVALUATE THE SAFETY AND EFFICACY OF LACOSAMIDE AS ADJUNCTIVE THERAPY IN JAPANESE AND CHINESE ADULTS WITH PARTIAL-ONSET SEIZURES WITH OR WITHOUT SECONDARY GENERALIZATION SAP/Amendment Number
Final SAP

Date

12 Sen 2

**Confidentiality Statement** 


Date Streether <12 Sep 2014>

12 Sep 2014>

This document cannot be used to support and the listed to support and the list This document is the property of UCB and may not – in full or in part – be passed on, reproduced, published, or otherwise used without the express permission of UCB.

> 

### STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

This document has been reviewed and approved per the Review and Approval of Clinical Documents Standard Operating Procedures. Signatures below indicate that the final version of the Statistical Analysis Plan (SAP) or amended SAP is released for execution.




## **TABLE OF CONTENTS**

| тт | TOE | ADDDEV | TATIONS | 1 | 5 |
|---|---|---|---|---|---|
| Lii<br>1 | | | IATIONSION | | |
| 2 | | | SUMMARY | | |
| <b>4</b> | 2.1 | | ojectives | | |
| | | | rimary objectives | | |
| | | | econdary objective | | 3.0 |
| | | Study ve | ariables | ~ | g.<br>6 |
| | 2.2 | Study va<br>1 Sa | afety variables | ~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~~ | 6 |
| | 2.2 | 2.1 50 | Primary safety variables Other safety variables Fricacy variables Primary efficacy variables Secondary efficacy variables Other efficacy variables esign and conduct nation of sample size YSIS CONSIDERATIONS presentation of summaries and analyses study level definition elative day nalysis time point ompleter cohort on of Baseline values | S10, | 6 |
| | | 2.2.1.1 | Other safety variables | 3 | 6 |
| | 2.0 | 2.2.1.2<br>2 Et | fficacy variables | , | 7 |
| | 2.2 | 2221 | Primary efficacy variables | , | ,<br>7 |
| | | 2.2.2.1 | Secondary efficacy variables | , | ,<br>7 |
| | | 2.2.2.3 | Other efficacy variables | , | ,<br>7 |
| | 2.3 | Study de | esign and conduct | , | ,<br>7 |
| | 2.4 | Determi | nation of sample size | 5 | 8 |
| 3 | DAT | A ANAL | YSIS CONSIDERATIONS - ** | ( | 9 |
| | 3.1 | General | presentation of summaries and analyses | ( | 9 |
| | 3.2 | General | study level definition | ( | 9 |
| | 3.2 | 2.1 R | elative day | ( | 9 |
| | 3.2 | 2.2 A | nalysis time point | ( | 9 |
| | 3.2 | 2.3 Co | ompleter cohort | 10 | 0 |
| | 3.3 | Definition | on of Baseline values | 10 | 0 |
| | 3.4 | | deviations | | |
| | 3.5 | | s sets | | |
| | 3.5 | | Il Subjects Screened | | |
| | 3.5 | | ifety Set | | |
| | 3.5 | | ıll Analysis Set | | |
| | 3.6 | Treatme | nt assignment and treatment group | 1 | 1 |
| | 3.7 | Center p | oooling strategy | 1 | 1 |
| | 3.8 | | dictionaries | | |
| 45 | | | L/ANALYTICAL ISSUES | | |
| | 4.1 | Adjustm | nents for covariates | 1 | 1 |
| | 4.2 | Handlin | g of dropouts or missing data | 1 | 1 |
| | 4.3 | Interim | analyses and data monitoring | 13 | 3 |
| | 4.4 | Multicer | nter studies | 13 | 3 |
| | 4.5 | Multiple | e comparisons/multiplicity | 13 | 3 |

| 3ep2014 |
|---------|
| EP0009 |

| | 4.6 | Use of an efficacy subset of subjects | 13 |
|---|---|---|---|
| | 4.7 | Examination of subgroups | 13 |
| 5 | STU | TDY POPULATION CHARACTERISTICS | 13 |
| | 5.1 | Subject disposition | 13 |
| | 5.2 | Protocol deviations | 14 |
| 6 | DEN | MOGRAPHICS AND OTHER BASELINE CHARACTERISTICS | 14 |
| | 6.1 | Demographics | 14\? |
| | 6.2 | Other Baseline characteristics | 4 |
| | 6.3 | Medical history and concomitant disease | |
| | 6.4 | Concomitant medications. | 15 |
| 7 | MEA | Demographics Other Baseline characteristics Medical history and concomitant disease Concomitant medications ASUREMENTS OF TREATMENT COMPLIANCE ETY ANALYSES Extent of exposure Adverse events Clinical laboratory evaluations Vital signs, physical findings, and other observations related to safety | 16 |
| 8 | SAF | ETY ANALYSES | 16 |
| | 8.1 | Extent of exposure | 16 |
| | 8.2 | Adverse events | 17 |
| | 8.3 | Clinical laboratory evaluations | 18 |
| | 8.4 | Vital signs, physical findings, and other observations related to safety | 19 |
| | 8. | 4.1 Vital signs | 19 |
| | 8. | 4.2 Electrocardiograms | 19 |
| | 8. | 4.1 Vital signs 4.2 Electrocardiograms 4.3 Other safety variables ICACY ANALYSES Statistical analysis of the primary officacy variables | 20 |
| 9 | EFF | ICACY ANALYSES | 21 |
| | 9.1 | Statistical analysis of the primary officacy variables | 21 |
| | 9.2 | Statistical analysis of the secondary efficacy variables | 21 |
| | 9.3 | Analysis of other efficacy variables | 22 |
| 10 | PHA | ARMACOKINETICS AND PHARMACODYNAMICS | 24 |
| 11 | OTF | IER ANALYSES | 24 |
| 12 | REF | ERENCES | 25 |
| 13 | APP | ENDICES | 26 |
| | 13.1 | List of Other Significant AEs | 26 |
| | 13.2 | Marked lab abnormalities | 28 |
| | | 3.2.1 Hematology | |
| | 13 | 32.2 Chemistry | 30 |
| | 13.3 | Vital sign assessments - abnormal | 33 |
| • | 13.4 | Electrocardiogram (ECG) – abnormal | |

### LIST OF ABBREVIATIONS

Analysis Set
Informed consent form
International League Against Epilepsy
Lacosamide
Lever function test
Iedical Dictionary for Regul
eferred term
ious adve
: Adverse event(s) AE(s) AED(s) **ALT AST** 

**CRF** ECG(s)

eCRF **EEG** 

**FAS** 

**ICF** 

**ILAE** 

**LCM** 

LFT

MedDRA

РТ

SAE(s)

QT interval corrected using Bazett's formula QTcB QT interval corrected using Fridericia's formula QTcF QT interval corrected using the population **QTcP** 

Statistical analysis plan SAP Standard deviation SD This document cannot be used to support amy System organ class SOC

Safety Set

Treatment-emergent adverse event

Upper limit of normal

World Health Organization Drug Dictionary


### INTRODUCTION

This Statistical Analysis Plan (SAP) describes the statistical principals that are applied for the This SAP should be read in conjunction with the following documents that provide all necessary background information and rationale for the current study and its design.

1) Finalized Study Protocol Amendment

2) Electronic Case P.

Lessa vertensions of val

#### 2 PROTOCOL SUMMARY

#### 2.1 Study objectives

#### 2.1.1 **Primary objectives**

The primary objectives of this study are the following:

- To evaluate the safety and tolerability of long-term administration of lacosamide (LCM) at doses up to 400mg/day in Japanese and Chinese adults with epilepsy who have completed the Treatment and Transition Period of EP0008
- To allow subjects who had completed the Treatment and Transition Periods of EP0008 to receive LCM

#### 2.1.2 Secondary objective

The secondary objective of this study is the following:

- To evaluate the efficacy of long-term administration of LCM at doses up to 400mg/day in Japanese and Chinese adults with epilepsy who have completed the Treatment and Transition Periods of EP0008
- 2.2 Study variables
- Safety variables 2.2.1

#### Primary safety variables 2.2.1.1

The primary safety variables are the following:

- Adverse events (AEs) reported spontaneously by the subject or observed by the investigator
- Subject withdrawals due to AEs

#### 2.2.1.2 Other safety variables

The other safety variables are the following:

- Changes in hematology, clinical chemistry, and urinalysis parameters
- Changes in 12-lead electrocardiograms (ECGs)
- Changes in vital sign measurements (ie, blood pressure, pulse rate)


Changes in body weight

#### 2.2.2 **Efficacy variables**

#### 2.2.2.1 Primary efficacy variables

No primary efficacy variables are defined for EP0009.

#### 2.2.2.2 Secondary efficacy variables

The secondary efficacy variables are the following:

- Percent change from Baseline in partial-onset seizure frequency per 28 days, where Baseline is defined as the Baseline Period of EP0008
- 50% response, where a responder is a subject experiencing a  $\geq$ 50% reduction from Baseline in partial-onset seizure frequency per 28 days, and Baseline is defined as the Baseline Period of EP0008

### 2.2.2.3

Other efficacy variables are the following:

- Other efficacy variables
  ner efficacy variables are the following:
  75% response, where a responder is a subject experiencing a ≥75% reduction from Baseline in partial-onset seizure frequency per 28 days and Baseline is defined as the Baseline Period of EP0008
- Subjects who achieved "seizure-free" status (yes/no)
- Percentage of seizure-free days
- Subjects who are changed to LCM monotherapy for at least 6 months
- Subjects who are changed to LCM monotherapy for at least 12 months

#### Study design and conduct 2.3

EP0009 is a Phase 3, multicenter, open-label, uncontrolled, extension study designed to evaluate the safety, tolerability, and efficacy of long-term administration of LCM as adjunctive therapy at doses up to 400mg/day in Japanese and Chinese adults with partial-onset seizures with or without secondary generalization who have completed the Treatment and Transition Periods of EP0008 and chose to enroll in EP0009.

Visit 1 of EP0009 is the same as the Final Visit of EP0008. Visits 2 through 4 of EP0009 will occur at 4-week intervals relative to the date of Visit 1. Beginning with Visit 5, each visit will occur at 12-week intervals relative to the date of Visit 1 until the End-of-Study/Withdrawal Visit.

At the completion of EP0008, all subjects who choose to enroll in EP0009 will be taking a dose of LCM 200mg/day. During the EP0009 Treatment Period, the investigator will be allowed to increase or decrease the doses of LCM and/or up to 3 concomitant antiepileptic drug(s) (AED[s]) to optimize tolerability and seizure reduction for each subject. The LCM dose may be decreased to 100mg/day or increased, no faster than 100mg/day per week, up to 400mg/day. Changes in concomitant AED(s) will be allowed only if the LCM dose has been stable for the previous 4 weeks; LCM dose must remain stable during changes to concomitant AED(s). Subjects may take no more than 3 concomitant AEDs except when temporary (≤12 weeks) use of an additional AED is required to switch to a new AED (ie, taper from old AED during titration of a new

 **UCB** 12Sep2014 Statistical Analysis Plan Lacosamide EP0009

AED). New AED(s) may be added only when the subject has not optimally or adequately responded to a maximum tolerated dose of LCM. The concomitant AED(s) can be carefully tapered or discontinued at the discretion of the investigator. Monotherapy with LCM is permitted. Increasing the dose of LCM and/or concomitant AED(s), as well as the addition of a new AED, should be done at a visit (scheduled or unscheduled).

At the end of the Treatment Period, an End-of-Study Visit will be required. If subjects prematurely withdraw from the study, a Withdrawal Visit will be required. Subjects who complete the Treatment Period and choose not to continue on to commercial LCM treatment, and subjects who prematurely withdraw from the study, will enter a Taper Period. During the Taper Period, subjects receiving doses greater than LCM 200mg/day at the End-of-Study/Withdrawal Visit should be tapered off gradually at a recommended decrease rate of LCM 200mg/day per week, unless the investigator feels that safety concerns require more rapid withdrawal of LCM. UCB (or designee) should be contacted if a more rapid withdrawal is required. A slower taper (e.g., LCM 100mg/day per week) is permitted, if medically necessary. Subjects receiving doses of LCM 200mg/day or lower at the End-of-Study/Withdrawal Visit are not required to taper off LCM. A Final Visit will be required 2 weeks after final LCM dose. Subjects who complete the Treatment Period and choose to continue on to commercial LCM treatment are not required to enter the Taper Period to taper off LCM or to return for a Final Visit; the End-of-Study Visit will be the last visit for these subjects. If LCM is not commercially available in a subject's country at the time the study closes, access to LCM will be provided according to local laws.

At selected sites, Japanese subjects may participate in an additional study (EP0024) with the intravenous formulation of LCM without withdrawing from EP0009. The study period of EP0024 will be included in that of EP0009. Subjects will continue to receive their current dose of LCM at the time of entry and remain stable for the duration of EP0024. Subjects who complete or withdraw from EP0024 will be given the opportunity to resume their participation in EP0009 with oral LCM treatment. In the event that a subject withdraws from EP0024 and is required to taper off LCM, the subject will return to EP0009 and taper using LCM tablets. Adverse events and concomitant treatment(s)/medication(s) that occur or were administered during EP0024 will be recorded in EP0024. Ongoing AEs and concomitant medication(s)/medical procedure(s) originating from the EP0024 will be followed in EP0009 until resolution or until stable. Where possible, data updates related to the resolution of ongoing AEs and concomitant medication(s)/medical procedure(s) from EP0024 will be reported in the EP0024 database (eg, updates are made in the EP0024 databases until the database is locked). All other data reported for EP0024 will be captured in the EP0024 database. Per the EP0024 protocol, the study (EP0024) will require hospitalization. Hospitalization for study participation does not need to be reported as an SAE.

### **Determination of sample size**

No formal sample size determination has been performed because EP0009 is an extension study. Approximately 378 subjects, ie, 70% of subjects who were randomized in EP0008, are anticipated to participate in this extension study.


12Sep2014 EP0009

### 3 DATA ANALYSIS CONSIDERATIONS

### 3.1 General presentation of summaries and analyses

Datasets will be analyzed using SAS version 9.1.3 or higher. All tables and listings will use Courier New font size 9.

Descriptive statistics will be displayed to provide an overview of the safety and efficacy results.

For categorical parameters, the number and percentages of subjects in each category will be presented at the relevant time point. The denominator for percentages will be based on the number of subjects appropriate for the purpose of analysis. Percentages will be presented to one decimal place. Percentages will not be presented for zero counts and 100% will be presented as an integer.

For continuous parameters, descriptive statistics will include number of the subjects, mean, standard deviation (SD), median, minimum, and maximum. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the CRF. The mean, SD, median will be reported to one more decimal place, than the raw data recorded in the CRF. In general, the maximum number of decimal places reported should be 4 for any summary statistics.

Subjects who withdraw early from the study will be evaluated based on the data collected at each visit attended or period entered. Data summaries will be presented overall and by randomized dose in EP0008 unless otherwise specified. Additionally, summaries will be presented separately by country.

### 3.2 General study level definition

### 3.2.1 Relative day

Relative day is defined as the day relative to the first dose in EP0009 of LCM.

- If the start date of an event occurred prior to the first dose of LCM in EP0009, the relative day is calculated as start date minus first LCM dose date. In subject data listings, relative days based on this situation will be preceded by a "-".
- If the start date of an event occurred on or after the first dose of LCM but prior to or on the last dose of LCM in EP0009, the relative day is calculated as start date minus first LCM dose date + 1.
- If the start date of an event occurred after the date of last dose of LCM in EP0009, the relative day is calculated as start date minus last dose date. In subject data listings, relative days based on this situation will be preceded by a "+".

### 3.2.2 Analysis time point

For analysis purposes, the Treatment Period is defined as the period of time from the first dose of study drug during the EP0009 study to the date of last dose of study drug or the date of ESV/WV, whichever occurs later. The Treatment Period includes time while treated with LCM during the protocol-defined Taper Period if the subject enters the Taper Period.

The Post-Treatment Period is defined as the treatment-free observational period after the Treatment Period. It starts one day after the end date of the Treatment Period and ends on the date of the final clinic visit or date of last contact with the subject, whichever is later. Data for


safety parameters evaluated at clinic visits (ie, laboratory, ECG, vital signs, weight, physical exam, and neurological exam) will be summarized for each visit during the Treatment Period. Additionally, the minimum and maximum values during the Treatment Period will be

Data from the Final Visit (2 weeks after final LCM dose) will be reported separately on by-visit summaries of safety parameters evaluated at clinic visits. It should be noted that all subjects available LCM do not require a Final Visit. Subjects completing the students available LCM do not require a Final Visit.

#### 3.2.3 **Completer cohort**

A completer cohort will be defined as the subset of subjects in the FAS that were enrolled and treated with LCM for a specified duration of time and have seizure diary data available for the duration of the cohort. For example, a 6-month completer cohort consists of subjects enrolled and treated with LCM for at least 6 months and have efficacy data through at least 1-year exposure where a month is defined as 28 days. EP0009 will last 3 years, so 6-month completer cohort, 12-month completer cohort, 18- month completer cohort, 24-month completer cohort, 30month completer cohort, and 36-month completer cohort will be defined in this study.

### **Definition of Baseline values** 3.3

Unless otherwise specified, Baseline will be defined from the Baseline values of EP0008and will be taken directly from EP0008 data sets (ie, not reprogrammed in EP0009).

For Baseline seizure frequencies, the partial-onset seizures per 28-days derived during the Baseline Period in EP0008 will be used. The number of lifetime AEDs from EP0008 and the number of concomitant AEDs taken during EP0008 will also be used.

For quantitative ECGs, Baseline was defined as the average of the 3 ECG measurements taken at Visit 3 of EP0008. If a subject had less than 3 ECG measurements on the day of Visit 3 of EP0008, Baseline was to be defined as the average of the available ECGs on the day of Visit 3 of EP0008. If no ECGs were available on the day of Visit 3 of EP0008, Baseline was not defined for ECG assessments.

For laboratory and vital sign data, Baseline was the last non-missing evaluation prior to the first dose of intake of the study drug in EP0008.

### Protocol deviations 3.4

The data will be reviewed to identify important protocol deviations. Important protocol deviations will be identified and documented prior to database snapshot for interim reports and database lock for the final analysis based on predefined criteria. Important deviations will be categorized as follows:

- Inclusion criteria
- Exclusion criteria
- Withdrawal criteria
- Prohibited medications
- Procedure non-compliance



12Sep2014 EP0009

### Other

A list of subjects with important protocol deviations will be agreed upon and documented prior to database lock.

All subjects Screened
All subjects screened will consist of all subjects who signed the informed consent form (ICF).

3.5.2 Safety Set
The Safety Set (SS) will include all enrolled and in EP0009.

#### 3.5.3 **Full Analysis Set**

The analysis set for the efficacy variables will be the Full Analysis Set (FAS) and will include all subjects in the SS having at least 1 day with available seizure diary data in EP0009.

#### Treatment assignment and treatment group 3.6

All subjects treated in EP0009 received LCM at doses ranging between 100mg/day to 400mg/day. A subject's LCM dose may be decreased to 100mg/day or increased, no faster than 100mg/day per week, up to 400mg/day. In terms of results presentation, summaries will present subjects overall and by randomized dose in EP0008: placebo, LCM 200mg/day, or LCM 400mg/day, unless otherwise specified.

#### Center pooling strategy 3.7

For the purpose of the summaries and analyses, the term 'Center' will be used to define each site.

All centers will be pooled by country for the purpose of analysis.

Descriptive summaries will not be presented by individual center. Subject data listing will provide data sorted by country and individual center.

#### 3.8 Coding dictionaries

All AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 16.1.

All medications will be coded using the World Health Organization Drug Dictionary (WHO-DD) version SEP/2013.

All coding will be performed prior to database lock.

### STATISTICAL/ANALYTICAL ISSUES

### Adjustments for covariates

This section is not applicable.

### Handling of dropouts or missing data

For by-visit analyses, data from the Withdrawal Visit will be presented with data corresponding to the next scheduled visit for the subject.

 Due to the potential for missing number of seizures for a given diary date, seizure frequency will be calculated using only the number of days for which seizure data is provided.

For analyses of treatment-emergent AEs (TEAEs) and concomitant medications, a complete date must be established in order to correctly identify the TEAE or medication as occurring during treatment or not. For purposes of imputing missing components of partially reported start and stop dates for adverse events and for medications, the algorithms listed below will be followed. Start and stop dates of AEs or concomitant medication will be displayed as reported in the subject data listings (ie, no imputed values will be displayed in data listing).

• Missing start day, but month and year present: If the start date of the data of the data and the same month and was present.

- Missing start day, but month and year present: If the start date of study treatment occurred in the same month and year as the occurrence of the event/medication, the start day of the event/concomitant medication will be assigned to the day of first intake of study treatment in order to treat the adverse event and medication as treatment-emergent and concomitant, respectively. Otherwise the start day will be set to the 1<sup>st</sup> day of the month?
- Missing start day and month, but year present: If the start date of trial medication occurred in the same year as the occurrence of the event/medication, the start day and month will be assigned to the date of first intake of study treatment in order to treat the adverse event and medication as treatment-emergent and concomitant, respectively. Otherwise the start day and month will be set to January 1<sup>st</sup>.
- Start date is completely unknown: The start date of the event/concomitant medication will be assigned to the date of first intake of study treatment.
- Missing end day, but month and year present: The end day will be set to the last day of the month.
- Missing end day and month, but year present: The end day and month will be set to the
  maximum of the date of study or the date equivalent to 30 days after last intake of study
  treatment.
- End date is completely unknown: The end date will not be imputed.

However, if the study termination year and year for the date which is 30 days after last intake of study treatment are greater than the event/concomitant medication year, the day and month are to be set to December 31<sup>st</sup>.

Relative day is not calculated for partial dates in cases where relative day is shown in a subject listing. In such cases, relative day should be left blank in the subject data listings.

Subjects participating in EP0024 while also enrolled in EP0009 will have missing data for seizure frequency and drug dosing while participating in the EP0024 trial. As the duration of the EP0024 study will be short (3-7 days), no imputation for data missing due to participation in EP0024 will be performed. Subjects will be assigned the same dose in EP0024 as that assigned in EP0009 for the two weeks prior to the start of EP0024. As such, time during the EP0024 study will not be subtracted from the exposure calculations (eg, exposure will be from the start of LCM treatment in the EP0009 study until the date of last dose of LCM in EP0009).

For the calculation of variables related to seizure frequency, the dates during participation in EP0024 will be considered as not done for the purpose of efficacy analyses for trial EP0009 (eg, these dates will not be considered as days evaluated for seizure frequency). Due to the short nature of the EP0024 study, only a few days of seizure frequency data are expected to be missing

12Sep2014 EP0009

due to participation in EP0024 unless otherwise specified (eg, for the evaluation of seizure freedom).

#### 4.3 Interim analyses and data monitoring

sudy to support regulatory submissions. At a minimum, 2 interim reports are planned after all enrolled Japanese subjects complete through Visit 5 (Week 24) and after all enrolled Japanese subjects complete through Visit 7 (Week 48). All analyses described in this SAP will be presented at each interim analysis for regulatory reporting

#### 4.4 **Multicenter studies**

Descriptive summaries for individual sites will not be presented due to the low number of expected subjects per site. However, subject data listings will provide data grouped by country and individual site.

#### 4.5 Multiple comparisons/multiplicity

This section is not applicable.

#### Use of an efficacy subset of subjects 4.6

Selected efficacy analyses will be performed for the completer cohorts defined in Section 3.2.3.

#### **Examination of subgroups** 4.7

Unless otherwise noted, all tabular data summaries will be presented overall and by country (Japan, China).

#### STUDY POPULATION CHARACTERISTICS 5

#### 5.1 Subject disposition

Summary tables of subject disposition will be provided overall, by EP0008 randomized dose and by country separately as follows:

- The number of subjects in the SS, and in the FAS will be presented. The date of the first visit for the first subject, date of the last visit for the last subject, and the number of subjects screened will also be included. (Analysis population: All Subjects Screened)
- The number and percentage of subjects entering, completing, ongoing, and discontinuing the study with associated reasons for discontinuation. The number and percentage of ongoing subjects will be displayed at the interim analyses only. (Analysis population: SS and FAS)
- A by-subject listing of analysis population classification (Analysis population: SS)

The following listing will be provided:

Subject disposition status, including the date of informed consent, screening result, date of study completing/discontinuation, and reason for premature discontinuation. (Analysis population: SS)

A by-subject listing of subjects who did not meet study eligibility criteria (Analysis population: All Subjects Screened)

 A by-subject listing of analysis population classification (Analysis population: SS)

#### 5.2 **Protocol deviations**

A summary table and listing of important protocol deviations will be provided for the SS as follows:

- The number and percentage of subjects with no important protocol deviations and with at least 1 important protocol deviation in each of the categories defined in Section 3.4 will be summarized overall, by EP0008 randomized treatment.
- A by-subject listing of important protocol deviations will be presented.

### 6 **DEMOGRAPHICS AND OTHER BASELINE CHARACTERISTICS**

Unless otherwise specified, demographics, baseline characteristics, medical history, concomitant disease, and concomitant medications will be summarized for the SS and FAS overall, by EP0008 randomized treatment group, and by country separately.

Subject listings of demographics, baseline characteristics, medical history, concomitant diseases, and concomitant medication will be displayed for the SS.

#### 6.1 **Demographics**

Summary statistics or the number and percentage for each category of demographic information will be presented as follows:

- A summary of demographics data including gender, age (years), age category ( $\leq 18$ , >18 to  $<65, \ge 65$  years) ( $<16, \ge 16$  to  $<65, \ge 65$  years), ethnicity (Hispanic or Latino, and not Hispanic or Latino), race group (American Indian/Alaskan native, Asian, Black, Native Hawaiian or other Pacific Islander, White, and Other/mixed), race, racial subgroup (Chinese or Japanese), height, weight, body mass index (BMI, kg/m<sup>2</sup>), BMI category (<18.5,  $\ge18.5$  to <25,  $\ge25$  to <30, and  $\ge 30 \text{ kg/m}^2$ ), number of lifetime AEDs, number of concomitant AEDs during EP0008, and Baseline partial-onset seizure frequencies per 28 days will be provided overall. by EP0008 randomized treatment group, and by country separately.
- A by-subject listing of demographic data.

Gender, race, ethnicity, racial subgroup, height, weight, and BMI will betaken directly from EP0008 datasets and not programmed. Age will be relative to the date of informed consent for EP0009.

### Other Baseline characteristics 6.2

Summary statistics or the number and percentage for each category of baseline characteristics as reported at Visit 1 of EP0008 will be provided as follows:

A summary of the diagnoses of primary disease, including time since diagnosis of epilepsy (in years) and etiology of epilepsy taken from EP0008 will be provided.

In EP0008, time since first diagnosis was calculated using all available information; partial dates was completed using the earliest calendar date based on the partial date provided.

 In EP0008, time since the first diagnosis (years) was calculated as (year and month of informed consent date – year and month of the first diagnosis) / 365.25. Month and year of the first epilepsy diagnosis are collected on the CRF. To calculate the time since first epilepsy diagnosis at Visit 1 of EP0008, a complete date will be imputed as follows:

- Missing the month, but year present assign January 1st of the year, the subject's birthday, or the date birthday, or the date of the first seizure, whichever is later in the year. Both month and year are missing, no imputation will be a subject of the year.
- A summary of International League Against Epilepsy (ILAE) seizure classification will be provided.

The types of partial seizures experienced will be summarized using the ILAE classification system.

- A summary of classification of epileptic syndromes.
- A by-subject listing of other Baseline characteristics.

#### 6.3 Medical history and concomitant disease

Medical history and concomitant diseases will be as reported as of Visit 1 of EP0008.

Concomitant diseases are medical history events which were ongoing at Visit 1 of EP0008.

Summary tables of medical history and concomitant diseases will be provided for the SS as follows:

- A summary of medical history by MedDRA system organ class (SOC) and preferred term (PT) will be presented overall, by EP0008 randomized treatment group, and country separately.
- A summary of concomitant disease by MedDRA system organ class (SOC) and preferred term (PT) will be presented overall, by EP0008 randomized treatment group, and country separately.
- A by-subject listing of medical history.
- A by-subject listing of concomitant diseases.
- A by-subject listing of procedure history.

## **Concomitant medications**

Concomitant medications will be defined as any medications taken concurrent with LCM if the start date was prior to the first dose with ongoing status, or the start date was on or after the date of first dose of study drug in EP0009. Medications with a missing start date, whose stop date is either unknown or after the date of the first dose of study drug, will be considered concomitant.

Summary tables will be provided for the SS and FAS as follows:

A summary of concomitant medications (excluding AEDs) taken during Treatment Period will be provided by level 1 and level 2 ATC code. The tables will be presented overall, by EP0008 randomized treatment group, and by country separately.


- A summary of concomitant AEDs taken during the Treatment Period will be provided by Level 4 ATC code and preferred medication name. The tables will be presented overall, by EP0008 randomized treatment group, and by country separately.
- A by-subject listing of concomitant AEDs (Analysis population: SS)
- A by-subject listing of concomitant medications (non-AEDs) (Analysis population: SS)

#### 7 MEASUREMENTS OF TREATMENT COMPLIANCE

LCM dosing compliance will be evaluated through the review of important protocol deviations classified under LCM Dosing Regimen.

### **SAFETY ANALYSES**

All safety analyses will be performed on the SS.

#### 8.1 **Extent of exposure**

Overall exposure to LCM in days is calculated as the date of last administration of LCM minus the date of first administration in EP0009 plus 1. Subject-years of exposure will be calculated as the number of days of exposure, divided by 365.25. Gaps in LCM treatment or days on the LCM dosing log CRF with unknown dosing will not be subtracted from the overall exposure days and subject-years of exposure.

The maximum daily dose will be calculated as the highest total daily dose the subject received during the treatment period.

LCM modal dose (mg/day) will be defined as the daily LCM dose the subject received for the longest duration during the treatment period in EP0009. A modal dose calculated as 50mg/day will be presented with 100mg/day. For any modal dose greater than 100mg/day falling between 2 consecutive categories, the modal dose will be presented with the lower of the consecutive categories. For example, 150mg/day will be presented with the 100mg/day group. The modal dose calculation is based on the number of days a subject was on a given daily dose. Gaps in LCM dosing will be excluded from the determination of modal dose (ie, no imputation for days with missing dosing log information will be performed).

The following exposure summaries and a listing will be produced:

- Summary statistics for study treatment duration (days) by modal dose and overall.
- Number of subjects and subject-years of study treatment duration by cumulative time intervals (ie, >0, >6, >12, >18, >24, >30, and >36 months, where one month is defined as 28
- dose, maximum daily dose, and overall. LCM treatment duration categories (days) are as follows: 1 to 14; 15 to 28; 29 to 56; 57 to 84; 85 to 168; 169to 336; 337 to 672. 673 to 1009 to 1344; 1345 to 1680; 1681 to 2016; ≥2017. any duration categories (days) are as some month is defined as Number and percentage of subjects within each LCM treatment duration category by modal follows: 1 to 14; 15 to 28; 29 to 56; 57 to 84; 85 to 168; 169to 336; 337 to 672; 673 to 1008;
  - maximum daily dose (mg/day) will be presented by EP0008 randomized treatment group and overall.

• A by-subject listing of LCM dosing.

#### 8.2 Adverse events

TEAEs will be coded using MedDRA and tabulated by SOC and PT. All summaries will be sorted alphabetically by SOC and by frequency of events in the overall column within the starting with the most frequent event unless otherwise specified.

The following summaries.

treatment group, and by country separately. For the summary tables of TEAEs onset during the Treatment Period will be further presented overall, by 6month interval, by EP0008 randomized treatment group, by country, and follows as well:

- Overview summaries of TEAEs with onset during the Treatment Period and events during the Post-Treatment Period will be presented. They will include the number and percentage of subjects with at least 1 TEAE, at least 1 serious TEAE, at least 1 TEAE leading to early withdrawal, drug-related TEAEs, at least 1 severe TEAE, and death.
- Summary of the incidence of TEAEs with onset during the Treatment Period by SOC and PT.
- Summary of the incidence of TEAEs with onset during the Treatment Period by SOC, PT, and maximum intensity.
- Summary of the incidence of TEAEs with onset during the Treatment by SOC, PT, and relationship.
- Summary of the incidence of serious TEAEs with onset during the Treatment by SOC and PT.
- Summary of the incidence of non-serious TEAEs by SOC and PT. The occurrence of nonserious TEAEs is only presented with incidence  $\geq 5\%$ .
- Summary of the incidence of TEAEs leading to discontinuation with onset during the Treatment Period by SOC and PT.
- Summary of the incidence of other significant TEAEs (Section 13.1) with onset during the Treatment Period by SOC and PT.
- Summary of incidence of TEAEs with onset during the Treatment Period per 100 personmonths of exposure.
- A sumi Périod.
  A sumi Périod. Assummary of subject numbers of subjects with TEAEs with an onset during the Treatment
  - A summary of subject numbers of serious TEAEs with an onset during the Treatment Period.
  - A summary of subject numbers of TEAEs with an onset during the Treatment Period leading to discontinuation.
  - A by-subject listing of all TEAEs; events with onset during the Post-Treatment Period will be identified.


- A by-subject listing for all deaths
- Glossary of MedDRA terms and associated investigator's terms for adverse events.

### 8.3 Clinical laboratory evaluations

For continuous laboratory measurements, including hematology, clinical chemistry, and urinalysis, a summary using descriptive statistics of the actual values and their change from Baseline (where Baseline is from the previous trial as defined in Section 3.3) will be presented at each visit, the last visit value, the minimum value, and the maximum value during the Treatment Period. For white blood cell differentials, both of absolute values and percentages of the white blood cell count will be analyzed. When analyzing categorical data, the number and percentage of subjects in each category will be presented. In addition, shift tables will be used to evaluate the number and percentage of subjects having a different Treatment Period status (low, normal, and high) when compared to their baseline status from EP0008.

Repeated or unscheduled laboratory assessments during the study will not be presented for each visit summary, but will be considered when determining the last visit value, minimum value, and maximum value during the Treatment Period and when determining treatment emergent marked abnormality.

Categorical urinalysis parameters (excluding urine glucose, urine ketones, and urine protein) will be presented in listings only.

The number and percentage of subjects with treatment-emergent marked laboratory abnormalities (hematology and clinical chemistry) as defined in Section 13 will be summarized by laboratory parameters. Treatment-emergent is defined as meeting the marked abnormality criteria during EP0009 Treatment Period but not meeting the criteria during Baseline of EP0008. Subject numbers for subjects meeting the marked abnormality criteria will also be presented.

A subject data listing will be provided for all laboratory data. Values outside the normal range will be flagged within the listing. A subject data listing will also be provided for all treatment-emergent marked laboratory abnormalities and will include all lab values for those subjects experiencing the marked abnormality.

The following summaries and listings will be provided:

- A summary of each laboratory parameter and change from Baseline of EP0008.
- A shift table based on the normal range for each lab parameter will be presented by Treatment Period endpoint value relative to Baseline of EP0008.
- A summary of incidence of treatment-emergent marked abnormalities presented by scheduled visit and for the entire Treatment Period (including unscheduled visits) during the Treatment Period for the laboratory parameters, hematology and clinical chemistry.

A shift table that will cross-tabulate Baseline value of EP0008 by maximum value during the Treatment Period (including unscheduled visits) will be presented for liver function tests (LFTs) which include alanine aminotransferase (ALT), aspartate aminotransferase (AST), GGT, ATL, and total bilirubin based on abnormality.


The shift table that cross-tabulates Baseline versus maximum values during the Treatment Period in categories of <1 x ULN, 1 to <2 x ULN, 2 to <3 x ULN, ≥3 x ULN, and missing will be presented for the liver function tests.

The summaries above will be provided overall, by EP0008 randomized treatment group, and by country separately.

• A by-subject listing of subjects with laborators.

- A by-subject listing of LFTs with pre-defined criteria.

### Vital signs, physical findings, and other observations related to 8.4 safety

#### Vital signs 8.4.1

Noninvasive pulse rate, systolic blood pressure, and diastolic blood pressure will be measured at visits with the subject in a sitting position after at least 3 minutes at rest, according to the tabular schedule of study procedures in the protocol. Summary statistics of the actual measurement and their changes from Baseline will be presented at each visit, the last visit value, the minimum value, and the maximum value during the Treatment Period

Repeated or unscheduled vital sign assessments during the study will not be presented for each visit summary, but will be considered when determining the last visit value, minimum value, and maximum value during the Treatment Period and post-Baseline abnormal vital signs during Treatment Period.

The following summaries and a listing will be provided:

- A summary of observed blood pressure and pulse rates and changes from Baseline of EP0008.
- The number and percentage of subjects with post-Baseline abnormal vital signs during Treatment Period as defined in Section 13.

The summaries above will be provided overall, by EP0008 treatment group, and by country separately.

A by-subject listing of vital signs. Abnormal vital signs will be flagged in the listing.

#### 8.4.2 Electrocardiograms

For quantitative ECG measurements (heart rate, RR interval, PR interval, QRS duration, QT interval, and corrected OT intervals using Bazett and Fridericia methods), summary statistics of the actual measurement collected at Baseline and each Treatment Period visit (as well as change from Baseline) will be presented. Baseline is defined as the average of the 3 ECG measurements taken at Visit 3 in EP0008. In addition to Baseline and each Treatment Period visit, the last visit, minimum, and maximum values during the Treatment Period of EP0009 will be presented. Repeated or unscheduled ECG assessments during the study will not be presented for each visit summaries, but will be considered when determining the last visit value, minimum value, and maximum value during the Treatment Period and abnormal ECG values.

The Bazett corrected QT (QTcB) will be calculated as

QTcB = 
$$\frac{QT}{\sqrt{RR}}$$
, where RR = 60/HR.

The Fridericia corrected QT (QTcF) will be calculated as

$$QTcF = \frac{QT}{\sqrt[3]{RR}}$$
, where  $RR = 60/HR$ 

The following summaries and listings will be provided for the SS:

- A summary of ECG measurements (heart rate, RR interval, PR interval, QRS duration, QT interval, and corrected QT intervals using Bazett and Fridericia methods) and changes and Baseline of EP0008.

  The number and percentage of and or
- and an increase from Baseline of <30ms, 30 to <60ms, and ≥60ms will be summarized for each visit.
- The number and percentage of subjects with a maximum QTc of 500ms, a maximum increase in QTc from Baseline of <30ms, 30 to <60ms, and ≥60ms, a maximum post-Baseline OTc of >500ms or a maximum increase in OTc of >60ms, and a maximum post-Baseline QTc of ≥500ms and a maximum increase in QTc of ≥60ms will be summarized for each of the corrected QT interval formulas. Subjects with a QTc (Bazett and Fridericia) of ≥500ms or an increase from Baseline of ≥60ms will be listed.
- The number and percentage of subjects with PR interval values >200ms, >220ms, or >250ms, and the number and percentage of subjects with ORS interval values >100ms, >120ms, and >140ms will be presented. For these defined criteria, the number and percentage of subjects with treatment-emergent PR interval and/or QRS interval prolongation will also be presented. Treatment-emergent is defined as meeting the criteria at any Treatment Period visit (including unscheduled visits) during the Treatment Period and not meeting the same criteria during Baseline.
- Subject numbers for subjects with prolonged post-Baseline QTcB will be provided.
- Subject numbers for subjects with treatment-emergent PR interval prolongation will be provided.
- Subject numbers for subjects with treatment-emergent QRS interval prolongation will be provided.
- A summary of incidence of treatment-emergent abnormality 12-lead ECG findings after start of study drug for each visit and during the Treatment Period in EP0009.

The summaries above will be provided overall, by EP0008 randomized treatment group, and by country separately.

- A by-subject listing of 12-lead ECG data.
- A by-subject listing of abnormal 12-lead ECG data as defined in Section 13.

#### 8.4.3 Other safety variables

Body weight will be determined without shoes when the subject is wearing light clothing, and will be assessed according to the tabular schedule of study procedures.

The following summaries and listings will be provided:

- A summary of body weight and change from Baseline for each visit

the Treatment Period as defined in Section 13.

The summaries above will be provided overall, by EP0008 randomized treatment group, and by country separately.

• A subject listing of body weight and change from Baseline in body weight

• A subject listing of abnormal physical examination abnormalities

• A subject listing of neurological examination findings

• A subject listing of pregnancy test

• A subject listing of C-SSRS suicidality

9 EFFICACY ANALYSES

All efficacy variables are to be evaluated descriptively using FASION

9.1 Statistical analysis of the primary efficacy variables.

No primary efficacy variables are defined for EP0009.

#### Statistical analysis of the secondary efficacy variables 9.2

Partial-onset seizure frequency per 28 days will be calculated as ([number of seizures over the specified interval] divided by [number of days in the interval]) multiplied by 28.

The following table and listing will be provided:

If a seizure cluster is reported, it will be assigned to the correct seizure type and the highest recorded daily number of seizures of that seizure type during the 28 days prior to the cluster event will be used as the imputed number of seizures for the day on which the cluster occurred. If no other seizures are recorded for that seizure type for the subject in the 28 days prior to the cluster event, the frequency will be set to 1 or the number of cluster episodes reported if more than 1 cluster event occurred on the same day.

### 9.2.1 Percent change in seizure frequency from Baseline to the Treatment Period

The percent change in partial-onset seizure frequency per 28 days from Baseline to the Treatment Period in 6-month interval is calculated by the following formula:

[(Seizure frequency per 28 days in 6-month interval during the Treatment Period) -(Seizure frequency per 28 days during Baseline Period)] x 100 (Seizure frequency per 28 days during Baseline Period)


Descriptive statistics will be calculated for the percent change in partial-onset seizure frequency per 28 days from Baseline to the Treatment Period in 6-month specified interval during the Treatment Period, and overall.

The percent change in 28-day seizure frequency per 28 days from Baseline among each completer cohort will also be displayed. A subject must have been treated with LCM and have available seizure diary data for the interval for each interval (eg, 6-month completer cohort subjects must be enrolled and taking trial medication for at least 6 months and have available seizure diary data for the interval) to be included in the 6-month completer cohort (see Section 3.2.3 for definition of completer cohort).

- A summary of the percent change in partial-onset seizure frequency per 28 days from Baseline will be presented by 6-month interval and overall Treatment Period.
- A summary of the percent change in partial-onset seizure frequency per 28 days from Baseline among each complete cohort will be presented. For each completer cohort, the percent change in 28-day seizure frequency per 28 days from Baseline will be presented by 6-month time interval..

The summaries above will be provided overall, by EP0008 randomized treatment group, and by country separately.

• A by-subject listing of number of seizure, seizure frequency per 28 days and percent change from Baseline by 6-month interval and overall Treatment Period.

# 9.2.2 Response to treatment of at least 50% from Baseline to the Treatment Period

 $\geq$ 50% responders are defined as subjects who experience a  $\geq$ 50% reduction in partial-onset seizure frequency per 28 days from Baseline to the 6-month interval or the Treatment Period which is defined at Section 9.2.1.

- The number and percentage of \$50% responders in the partial-onset seizure frequency per 28 days from Baseline to the Treatment Period by 6-month interval and overall Treatment Period will be presented.
- The number and percentage of  $\geq 50\%$  responders among each completer cohort will be presented in a same way as above. For each completer cohort, the  $\geq 50\%$  response rate will be presented by 6-month time interval.

The summaries above will be provided overall, by EP0008 randomized treatment group, and by country separately.

• A by-subject listing of ≥50% responder categories by 6-month interval and overall Treatment Period.

### 93 Analysis of other efficacy variables

# 9.3.1 Response to treatment of at least 75% from Baseline to the Treatment Period

 $\geq$ 75% responders are defined as subjects who experience a  $\geq$ 75% reduction of in the partial-onset seizure frequency per 28 days from Baseline to the 6-month time interval or the Treatment Period.


- ≥75% responders will also be summarized by the same manner as ≥50% responders, described in Section 9.2.2.
- The number and percentage of ≥75% responders in the partial-onset seizure frequency per 28 days from Baseline to the Treatment Period by 6-month interval and overall Treatment Period will be presented.
- The number and percentage of  $\geq$ 75% responders among each completer cohort will be presented in a same way as above.

The summaries above will be provided overall, by EP0008 randomized treatment group, and by country separately.

• A by-subject listing of ≥75% responder categories by 6-month interval and overall Treatment Period.

### 9.3.2 Seizure-free status

A seizure-free status will be assessed for the duration of at least consecutive 6 months (182 days) and at least consecutive 12 months (365 days). Seizure-free is defined as a report of no seizures in the seizure diary on the CRF for the consecutive days where the subject was treated with LCM. Days in the seizure diary which are marked as "not done" on the CRF will not be counted as a seizure free day unless otherwise noted.

When subjects are in EP0024, the days should be treated as "not done" days for EP0009 but they should not disqualify a subject from being seizure free if they were in EP0024.

- The number and percentage of subjects who achieved seizure-free status (yes/no) for the duration of at least 6 months and at least 12 months will be presented overall, by completer cohort, by EP0008 randomized treatment group, and by country separately.
- A by-subject listing of seizure freedom data.

### 9.3.3 Percentage of seizure-free days

Percentage of seizure-free days is calculated as:

Seizure free days during time interval in the Treatment  $\frac{\text{Percentage of seizure free days}}{\text{Seizure free days}} = \frac{\frac{\text{Period}}{\text{Number of days during time interval in the Treatment}}}{\text{Number of days during time interval in the Treatment}} \times 100\%$ 

Time interval is defined as 6-month interval for the first year and yearly intervals thereafter (at least 6 months, at least 12 months, at least 24, and at least 36 months).

- Summaries of the percentage of seizure-free days during the Treatment Period will be presented overall, by completer cohorts, EP0008 randomized treatment group, and by country separately.
- A summary of change in percentage of seizure-free days and change in percentage from Baseline from Baseline during the Treatment Period will be presented overall, by completer cohorts, by EP0008 randomized treatment group, and by country separately.

#### 9.3.4 Subjects receiving LCM as monotherapy

Monotherapy is defined as when LCM only is used during the period with no other concomitant AEDs. If the subjects had a rescue medications of benzodiazepines which are used for the control of uncountable seizures due to clustering are not regarded as AEDs. Other AED rescues where an AED was taken for ≤1 day will also not disquality a subject from being on LCM monotherapy.

The number and percentage of subjects achieving continuous LCM monotherapy for at least 6 months and at least 12 months at any time during the Treatment Period among subjects who were exposed to LCM for at least 6 months and at least 12 months are least 12 months and at least 12 months are least 12 months and at least 12 months and at least 12 months are least 12 months and at least 12 months and at least 12 months are least 12 months and at least 12 months are least 12 months at least 12 months are least 12 months and at least 12 months are least 12 months at least 12 months are leas ACODYN,

ACODYN,

ACODYN,

ACODYN,

ARABITA AR

### PHARMACOKINETICS AND PHARMACODYNAMICS

The document control he used to support any materials altered to the support of t


## 13 APPENDICES

## 13.1 List of Other Significant AEs

| MedDRA Preferred Term |
|---|
| HEPATOTOXICITY RELATED TERMS |
| Hepatitis toxic |
| Hepatotoxicity |
| CARDIAC AND ECG RELATED TERMS |
| Atrioventricular block third degree Atrioventricular block second degree |
| Atrioventricular block second degree |
| Atrioventricular block second degree Bradyarrhythmia* |
| Bradycardia* |
| Bradycardia* Cardiac pacemaker insertion Atrial fibrillation Atrial flutter Sinus bradycardia* |
| Atrial fibrillation |
| Atrial flutter |
| Sinus bradycardia* |
| Ventricular tachycardia |
| Ventricular fibrillation |
| Heart Rate decreased* |
| Sick sinus syndrome |
| SUICIDALITY RELATED TERMS |
| Completed suicide |
| Depression suicidal |
| Suicidal behaviour |
| Suicidal ideation |


| | MedDRA Preferred Term | |
|---|---|---|
| Suicide attempt Intentional self-injury Self injurious behaviour Self-injurious ideation Intentional overdose Multiple drug overdose intentional Poisoning deliberate ADDITIONAL TERMS Loss of consciousness Syncope | | |
| | Intentional self-injury | |
| | Self injurious behaviour | |
| | Self-injurious ideation | of value |
| | Intentional overdose | ational and heart rate will be reviewed and only cases with marked bradycardia by with HR <45 bpm will be listed as 'Other Significant AEs'. A day that the lift of the listed as 'Other Significant AEs'. |
| | Intentional self-injury Self injurious behaviour | tells |
| | Poisoning deliberate | and |
| | ADDITIONAL TERMS | n ano |
| | Loss of consciousness | licatio. |
| | Syncope | ORT ARRY |
| This doc | unent cannot be used to support any marketing at | |


### 13.2 Marked lab abnormalities

### 13.2.1 Hematology

Abnormality criteria to be applied in the assessment of laboratory parameter values are given below.

| PARAMETER | AGE<br>RANGE | UNIT (conventional) | ABNORMALITY<br>CRITERIA | UNIT<br>(standard) | ABNORMALITY<br>CRITERIA |
|---|---|---|---|---|---|
| | | | (conventional<br>unit) | | (standard unit) |
| Hematocrit | <2y | % | ≤27<br>>45 | % | <u>≤27</u><br>≤107 >45 |
| | 2y -<br><17y | | ≤29<br>>47 | Sally of | ≤29<br>>47 |
| | ≥17y | | ≤85% of LLN<br>≥115% of ULN | 1/1- | |
| Hemoglobin | <2y | g/dL | ≤9.0<br>>15.0 | o g/L | ≤90<br>>150 |
| | 2y -<br><17y | | ≤9.5<br>≥16.0 | | ≤95<br>>160 |
| | ≥17y | | ≤85% of LLN<br>≥115% of ULN | | ≤85% of LLN<br>≥115% of ULN |
| WBC/Leukocytes | All | 10 <sup>9</sup> /L | ≤3.0<br>≥16.0 | G/L | ≤3.0<br>≥16.0 |
| Lymphocytes<br>Absolute | <2y | 10°/LOP | <1.0<br>>9.8 | G/L | <1.0<br>>9.8 |
| | 2y - <6y | aikeill | <0.7<br>>6.9 | | <0.7<br>>6.9 |
| | ≥6y | SUA LUG | <0.6<br>>5.0 | | <0.6<br>>5.0 |
| Basophils | >1m | % | ≥5.0 | % | ≥5.0 |
| Basophils<br>Absolute | >lm | 10 <sup>9</sup> /L | ≥0.4 | G/L | ≥0.4 |
| Eosinophils | >1m | % | ≥10 | % | ≥10 |
| Eosinophils<br>Absolute | >1m | 10 <sup>9</sup> /L | ≥1.0 | G/L | ≥1.0 |
| Monocytes | >1m | % | ≥20.0 | % | ≥20.0 |
| Monocytes<br>Absolute | >1m | 10 <sup>9</sup> /L | ≥2.0 | G/L | ≥2.0 |
| Neutrophils<br>Absolute | >1m | 10 <sup>9</sup> /L | <1.5 | G/L | <1.5 |
| Platelets | >1m | 10 <sup>9</sup> /L | ≤100<br>≥600 | G/L | ≤100<br>≥600 |


| <3.0 |
|--------------------------------------------|
| <3.5 × |
| Vallati |
| or 10 |


### 13.2.2 Chemistry

Abnormality criteria to be applied in the assessment of chemistry parameter values are given below.

| <b>PARAMETER</b> | AGE | UNIT | ABNORMALITY | UNIT | ABNORMALITY |
|---|---|---|---|---|---|
| | RANGE | (conventional) | CRITERIA | (standard) | CDITEDIA |
| | | (************************************** | (conventional) | ( | (standard) |
| AST (SGOT) | All | U/L | ≥3.0 x ULN | U/L | ≥3.0 x ULN |
| | | | ≥5.0 x ULN | | ≥5.0 x ULN |
| | | | ≥10.0 x ULN | | ≥10.0 x ULN |
| ALT (SGPT) | All | U/L | ≥3.0 x ULN | U/L | ≥3.0 x ULN |
| | | | ≥5.0 x ULN | | ≥5.0 x ULN |
| | | | ≥10.0 x ULN | U/Lyet | ≥10.0 x ULN |
| Alkaline | <4y | U/L | ≥690 | U/L O | ≥690 |
| Phosphatase | 4 | | . 024 | 'SIL'S | . 024 |
| | 4y - | | ≥834 | allo | ≥834 |
| | <10y | | > 17/(1 | 00.0 | > 177.1 |
| | 10y - | | ≥1761 | | ≥1761 |
| | <17y | | ijO | | ≥3.0 x ULN |
| | ≥17y | | ≥3.0 x ULN | | ≥3.0 X ULN |
| GGT | <6m | U/L | ≥522 | U/L | ≥522 |
| | ( ,1 | ć | | | > 270 |
| | 6m - <1y | ort any marketing | 21th <sup>O</sup> ≥279 | | ≥279 |
| | 1y - | 8-11-10° | ≥66 | | ≥66 |
| | <13y | Heil | 10.5 | | |
| | 13y - | Wal. | ≥126 | | ≥126 |
| | <17y | .d | >20 HIN | | >20 11131 |
| | ≥17y | A DIVI | ≥3.0 x ULN | | ≥3.0 x ULN |
| Total Bilirubin | >1m | mg/dL | ≥2.0 | umol/L | ≥34.208 |
| | 30 | | | | |
| Total Protein | 2m-<1y | g/dL | <3.0 | g/L | <30 |
| | 60 | | >11.9 | | >119 |
| A Marinot De | 1y - | | <4.3 | | <43 |
| 0,70 | <17y | | >12.0 | | >120 |
| anine | ≥17y | | <4.3 | | <43 |
| A 11 | z1 | - / JT | >13.0 | - /T | >130 |
| 1 Adminin | <1y | g/dL | <1.6<br>>7.2 | g/L | <16<br>>72 |
| Acciline min | >1177 | | >7.2<br><2.4 | | >72<br><24 |
| 40 | ≥1y -<br><17y | | >8.4 | | >84 |
| | ≥17y | | <2.6 | | <26 |
| | _1 / y | | ~2.0 | | ~20 |
| | l | l | I | | 1 |


| PARAMETER | AGE | UNIT | ABNORMALITY | UNIT | ABNORMALITY |
|---|---|---|---|---|---|
| | RANGE | (conventional) | CRITERIA | (standard) | CRITERIA |
| DADA | | / 17 | (conventional) | 1/7 | (standard) |
| BUN | <1y | mg/dL | ≥24 | mmol/L | ≥8.568 |
| | 1y - | | ≥36 | | ≥12.852 |
| | <17y | | | | ion |
| | ≥17y | | ≥40 | | ≥14.28 |
| Urea | <1y | mg/dL | >42 | mmol/L | >7.014 |
| | ≥1y | | >60 | | >10.02 |
| Creatinine | 1y - | mg/dL | >1.2 | umol/L | >106.8 |
| | <10y | | | ally | |
| | 10y -<br><16y | | >1.8 | umol/Lef | >159.12 |
| | ≥16y | | ≥2.0 | 000 | ≥176.8 |
| Creatinine | All | mL/min | 50 RP | mL/s | <0.835 |
| Clearance* Bicarbonate | >1m - | mEa/I | \$15 | mmol/L | <15 |
| Dicar voltate | <17y | mEq/L | ₹P : 1238 | IIIIIIOI/L | >38 |
| | ≥17y | Ć | ×18 | | <18 |
| | | 1.0K | >38 | | >38 |
| Calcium | <1y | mg/dl | < 6.9 | mmol/L | <1.725 |
| | | Leili | >12.2 | | >3.05 |
| | 1y - | adil | <7.4 | | <1.85 |
| | <17y | ation | >11.7 | | >2.925 |
| | ≥17y | mg/deketing | ≤7.6 | | ≤1.9 |
| C1.1 · 1 | . 1 | 001 | ≥11.0 | 1/7 | ≥2.75 |
| Chloride | >1m | mEq/L | ≤90<br>≥112 | mmol/L | ≤90<br>≥112 |
| D1 1 | | | ≥112 | 1/7 | ≥112 |
| Phosphorous | sly | mg/dL | <1.8 | mmol/L | <0.5814 |
| _ | . (3) | | >8.2 | | >2.6486 |
| . 0 | ly - | | <1.8 | | <0.5814 |
| Ol | <17y | | >7.4 | | >2.3902 |
| at cannot be | ≥17y | | ≤2.0 | | ≤0.646 |
| Potassium | z1 | 17 /1 | ≥6.0 | 1/T | ≥1.938 |
| Potassium | <1y | mEq/L | ≤3.0<br>≥6.5 | mmol/L | ≤3.0<br>≥6.5 |
| chi. | <u> </u> | | ≥6.5 | | ≥6.5 |
| 0 | ≥1y | | ≤3.0 | | ≤3.0 |
| G 1: | . 1 | T /T | ≥6.0 | 1 /w | ≥6.0 |
| Sodium | >1m | mEq/L | <127 | mmol/L | <127 |
| | | | >151 | | >151 |


| <b>PARAMETER</b> | AGE | UNIT | ABNORMALITY | UNIT | ABNORMALITY |
|---|---|---|---|---|---|
| | <i>RANGE</i> | (conventional) | CRITERIA | (standard) | CRITERIA |
| | | | (conventional) | , , | (standard) |
| Glucose | >1m - | mg/dL | < 50 | mmol/L | <2.775 |
| | <17y | | ≥180 | | ≥9.99 |
| | ≥17y | | < 50 | | <2.775 |
| | | | ≥200 | | ≥11.1 |
| Total | ≥1y | mg/dL | >250 | mmol/L | >6.475 |
| Cholesterol | | | | | 1,0, |
| LDL | 1y - | mg/dL | >140 | mmol/L | >3.626 |
| (calculated) | <17y | | | | ;ol <sup>2</sup> |
| | ≥17y | | >200 | × | >5.18 |
| HDL | ≤2y | mg/dL | <10 | mmol/L | < 0.259 |
| 1122 | | 1118, 4.2 | | any | 0.20 |
| | >2y | | <20 | mmol/Let | < 0.518 |
| | , | | | | |
| Triglycerides | <1y | mg/dL | >750 | o` mmol/L | >8.475 |
| | | | i Co | | |
| | ≥1y | | >300 | | >3.39 |
| ** * * * 1 | .4 | / 17 | 0,55 | 1 /7 | 455.006 |
| Uric Acid | <1y | mg/dL REDAC | ₹9.7 | umol/L | >457.996 |
| | 1y - | ć | >6.5 | | >386.62 |
| | <13y | OR | alili. V.S | | 300.02 |
| | 13y - | 24,00 | >8.6 | | >511.528 |
| | <17y | (etill) | | | |
| | ≥17y | Silk | >9.5 | | >565.06 |
| | | 141 | | | |
| Thyroxine (T4) | <1y | oug/dL | ≤4.3 | nmol/L | ≤55.3453 |
| | | OIL | ≥18.4 | | ≥236.8264 |
| | ≥1y | 8 | ≤3.8 | | ≤48.9098 |
| | 50 | • | ≥13.5 | | ≥173.7585 |
| Globulin | <1y | g/dL | <1.0 | g/L | <10 |
| | SO | | >4.5 | | >45 |
| ~° | ≥1y | | <1.2 | | <12 |
| X.V | | | >5.3 | | >53 |

ALT= alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen; dL = deciliter; GGT: gamma-glutamyltransferase; HDL = high density lipoprotein; LDL = low density

mpoprotein.

\*Schwartz equation (subjects <12): Cr Cl ml/min = [Height (cm) \* 0.55] / serum creatinine

Cockroft equation (subjects ≥12): Male: Cr Cl ml/min = [(140-age) x body weight (l/a)] / Cr

creatinine); Female: Cr Cl ml/min = [(140-age) x body weight (l/a)] / Cr Cockroft equation (subjects ≥12): Male: Cr Cl ml/min = [(140-age) x body weight (kg)] / (72 x serum creatinine); Female: Cr Cl ml/min =  $[(140\text{-age}) \times \text{body weight (kg)}] / (72 \times \text{serum creatinine})] \times 0.85$ 


## 13.3 Vital sign assessments - abnormal

Abnormality criteria to be applied in the assessment of vital signs parameter values are given below.

| ociow. | | |
|---|---|---|
| PARAMETER | AGE<br>RANGE | ABNORMALITY CRITERIA |
| Pulse Rate | <6m | <100 |
| (beats/minute) | | >180 |
| | 6m - <3y | <90 |
| | | >150 |
| | 3y - <12y | <u> </u> |
| | 3 y 12 y | <60<br>>130 |
| | 12y - <17y | <u>~</u> |
| | , , | ≤50<br>≥120 |
| | ≥17y | ≤50 and a decrease from Baseline of ≥15 |
| | | $\geq 120$ and an increase from Baseline of $\geq 15$ |
| Systolic Blood | <6m | <60 |
| Pressure (mmHg) | | . >100 |
| | 6m - <3y | . call < 70 |
| | , | >120 |
| | 3y - <12y | <80 |
| | | >140 |
| | 12y - <17y | <90 |
| | 129 179 | >160 |
| | ≥17y | ≥ 90 and a decrease from Baseline of ≥20 |
| | <u>-</u> 17 y | $\geq$ 180 and an increase from Baseline of $\geq$ 20 |
| Diastolic Blood | <6m | <40 |
| Pressure (mmHg) | om » | >65 |
| | 6m - <3y | <45 |
| | om 3/(, | <43<br>>75 |
| | 3y - <12y | |
| | 59 129 | <50<br>>80 |
| | 12y - <17y | |
| | S12y 117y | <u>&lt;50</u> |
| 7,60 | > 177 | >105 |
| used to | ≥17y | ≤50 and a decrease from Baseline of ≥15 |
| | | $\geq$ 105 and an increase from Baseline of $\geq$ 15 |
| Respiratory Rate | <6m | <25 |
| (breams/minute) | | >55 |
| Respiratory Rate (breaths/minute) | 6m - <3y | <20 |
| , ci | | >45 |
| Ve, | 3y - <12y | <15 |
| 3 | | >35 |
| | ≥12y | <10 |
| | | >25<br>>101 °F (38.3 °C) |
| Temperature | >1m | >101 °F (38.3 °C) |
| | 1 | |


## 13.4 Electrocardiogram (ECG) – abnormal

Abnormality criteria to be applied in the assessment of ECG parameter values are given below:

| Parameter | Age | Abnormality Criteria |
|---|---|---|
| QT interval (ms) | 1m-<12y | ≥500 |
| | ≥12y | ≥500 or ≥60ms increase from Baseline |
| QTc(F) (ms) | <6m | >490, or >15% increase from Baseline |
| | 6m-<3y | >440, or >15% increase from Baseline |
| | 3y-<12y | >440, or >15% increase from Baseline |
| | ≥12y- <17y | >440, or >15% increase from Baseline |
| | ≥17y | ≥500 or ≥60ms increase from Baseline |
| QTc(B) (ms) | <6m | >490, or >15% increase from Baseline |
| | 6m-<3y | >450, or >15% increase from Baseline |
| | 3y-<12y | >450, or >15% increase from Baseline |
| | ≥12y- <17y | >450, or >15% increase from Baseline |
| | ≥17y | ≥500 or ≥60ms increase from Baseline |
| PR interval (ms) | <6m | >150, or ≥25% increase from Baseline |
| | 6m-<3y | >170, or >25% increase from Baseline |
| | 3y-<12y | >180, or <u>&gt;</u> 25% increase from Baseline |
| | ≥12y - <17y | >200, or >25% increase from Baseline |
| | ≥17y | Treatment-emergent value >200, >220, >250 |
| QRS interval (ms) | €6m | >90, or ≥25% increase from Baseline |
| | 6m-<3y | >90, or ≥25% increase from Baseline |
| , 10 | 3y-<12y | >100, or <u>&gt;</u> 25% increase from Baseline |
| 1580 | ≥12y - <17y | ≥110, or ≥25% increase from Baseline |
| "PE" | ≥17y | Treatment-emergent value >100, >120, >140 |
| Heart rate (bpm) | <6m | <100,>180 |
| AT COST | 6m-<3y | <90,>150 |
| U.O. | 3y-<12y | <60,>130 |
| r | ≥12y | <50, >120 |

Note: Treatment-emergent is defined as meeting the criteria at any post-Baseline visit during the Treatment Period (including unscheduled visits) and not meeting the same criteria during Baseline

